CLINICAL TRIAL: NCT03680040
Title: Prospective Non-randomized Single Arm Multi-center Evaluation of the Durability of Aortic Bioprostheses/Valves With RESILIA Tissue in Subjects Under 65 (RESILIENCE Trial)
Brief Title: RESILIENCE Trial: Evaluation of the Durability of Aortic Bioprostheses/Valves With RESILIA Tissue in Subjects Under 65
Acronym: RESILIENCE
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-06
Record Dates: First submitted 2018-09-10; First posted 2018-09-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Subjects previously implanted with a RESILIA aortic tissue valve. — Subjects to undergo multi-slice computed tomography and echocardiogram to assess predictors of valve durability in previously implanted Edwards aortic valves with RESILIA tissue.

SUMMARY:
The objective of this observational trial is to determine time to valve failure due to valve deterioration requiring re-intervention and collect/investigate early potential predictors of valve durability (e.g., calcification and hemodynamic deterioration) in RESILIA tissue valves.

DETAILED DESCRIPTION:
Multicenter, prospective, non-randomized, single-arm, observational trial. Subjects will be evaluated at 5, 7, 9, and 11 years post-implant. Up to two hundred fifty (250) total subjects at up to fifteen (15) investigational sites will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Subject currently has an Edwards pericardial aortic bioprosthesis with RESILIA tissue
3. Provides voluntary written informed consent prior to the first trial related procedure
4. Subject agrees to attend follow-up assessments as specified in the protocol

Exclusion Criteria:

1. Age 65 years or older at time of aortic valve replacement
2. The Subject is pregnant or planning to become pregnant at the time of screening
3. Re-intervention required on the bioprosthetic aortic valve prior to screening
4. Active endocarditis or history of endocarditis on bioprosthetic aortic valve
5. Estimated life expectancy <24 months
6. Subjects with history of or current renal failure requiring dialysis
7. Altered mineral metabolism (hyperparathyroidism, parathyroid tumors)
8. Has prior organ transplant or is currently an organ transplant candidate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects previously implanted with a RESILIA aortic tissue valve.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Time to bioprosthetic valve failure due to valve deterioration | 11 years post-implant
  Time to bioprosthetic valve failure due to valve deterioration is defined as subject requiring valve re-intervention (redo surgery, valve-in-valve) or confirmed study valve-related death.

SECONDARY OUTCOMES:
Collection of early possible predictors of valve failure including leaflet calcification and morphological/hemodynamic valve deterioration | 5, 7, 9, and 11 years post-implant
  1. Quantification of valve leaflet calcification via core lab evaluated multi-slice computed tomography (MSCT)
  2. Hemodynamic performance of the valve and evaluation for possible morphological/hemodynamic valve deterioration confirmed by core lab evaluation of echo-cardiography

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bavaria, MD, Principal Investigator — Organizational Affiliation: Hospital of the University of Pennsylvania; Lars Svensson, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (10):
- United States (10):
  - University of Southern California, Los Angeles, California
  - University of Florida - Shands Hospital, Gainesville, Florida
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Columbia University Medical Center-NY Presbyterian Hospital, New York, New York
  - Weill Cornell - NYC, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pinnacle Health, Mechanicsburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine - St. Luke's Hospital, Houston, Texas
  - The Heart Hospital of Baylor Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.